CLINICAL TRIAL: NCT06185348
Title: Body Mass Index and Growth Parameters Evolution in Children Treated With Hybrid Closed Loop System for Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, RENARD Emeline, Doctor, Central Hospital, Nancy, France
Other Study IDs: 2023PI142
Record Dates: First submitted 2023-10-12; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 1; Obesity; Overweight; Child Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Obesity; Overweight; Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Overweigth and obesity are commonly diagnosed in children with type 1 diabetes, and frequently an increase of wiegth and BMI is observed after diagnoses. Hybrid cloosed loop system are new system where insulin is continually adapted to glycemia (using an algorythme). The weight and growth trajectory of children treated with this system is poorly described.

DETAILED DESCRIPTION:
Unlike type 2 diabetes, which is a frequent metabolic complication of obesity, type 1 diabetes is not a consequence of overweight or obesity, or of an excessively sweet or unbalanced diet.

However, more and more studies are linking type 1 diabetes to obesity. An international study with 23 026 children suffering from type 1 diabtes has shown that 22.3% of boys and 27.2% of children have overweight, and 6.8% and 6.3% respectively obesity . Several hypothesis are made to explain this trend : a consequence of intensive insulinotherapy, the fear of hypoglycemia with unnecessary glucose intake, the increase of caloric intake and the decrease of physcial activity. Moreover, subcutaneous insulinotherapy leads to modification in body composition with a increase in fat mass . Nevertheless, some studies highlights a possible role of obesity in the type 1 diabetes development( familial history of type 2 diabetes more common in children with type 1 diabetes , inverse relation with age at diagnosis and BMI suggesting that children with higher BMI will be diagnosed early in age .

Hybrid closed-loop systems, in which the insulin flow rate is adjusted almost instantaneously to the blood glucose level by using an algorithm with a CSII and a CGM, are new systems that have gradually been used in current practice . These systems are significantly associated with an improvement in glycemic control (HbA1C and TIR)[17], a reduction in the time spent in hypoglycemic states , and with an improvement in quality of life.

Nevertheless, the impact of this new treatment on weight evolution has been poorly described. A previous study with 50 children included did not show a BMI modification after 1 year of treatment. Individually, some patients following in our center have shown a reduction of BMI after treatment of type 1 diabetes with with hybrid closed loop system.

This leads us to perform an observational study in order to describe the trajectory of BMI and growth parameters of children suffering from type 1 diabetes (expressed in standard deviations (SDS) after 6 months, 1 year and 2 years of treatment with hybrid closed loop system in the university hospital of Nancy. The second objective is to identify potential factors associated with the positive evolution of BMI at 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* children between 6 and 18 years at the beginning of treatment with HCL
* type 1 diabetes
* follow up in University Hospital of Nancy between 01/01/2021 - 31/12/2023
* treatement with HCL since 6 months

Exclusion Criteria:

* parental opposition for the study
* pregnancy

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with type 1 diabetes follow up in Hospital of Nancy with HCL since 6 months minimum
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Body mass index (BMI) variation after 6 months of treatment with hybrid closed loop (HCL) | 6 months
  variation of BMI expressed in standard deviations after 6 months with HCL

SECONDARY OUTCOMES:
Body mass index (BMI) variation after 12 months of treatment with hybrid closed loop (HCL) | 12 months
  variation of BMI expressed in standard deviations after 12 months with HCL
Body mass index (BMI) variation after 24 months of treatment with hybrid closed loop (HCL) | 24 months
  variation of BMI expressed in standard deviations after 24 months with HCL
Growth velocity variation after 6 months of treatment with hybrid closed loop (HCL) | 6 months
  variation of Growth velocity expressed in standard deviations after 6 months with HCL
Growth velocity variation after 12 months of treatment with hybrid closed loop (HCL) | 12 months
  variation of Growth velocity expressed in standard deviations after 12 months with HCL
Growth velocity variation after 24 months of treatment with hybrid closed loop (HCL) | 24 months
  variation of Growth velocity expressed in standard deviations after 24 months with HCL
description of metabolic parameters at 6 months | 6 months
  HbA1C at 6 months
description of metabolic parameters at 12 months | 12 months
  HbA1C at 12 months
description of metabolic parameters at 24 months | 24 months
  HbA1C at 24months

IPD SHARING:
Plan to Share IPD: No